CLINICAL TRIAL: NCT02168998
Title: Level of Cortisol in Stress Response During Intravenous Access in the Pediatric Emergency Department With a Medical Clown: a Randomized Prospective Pilot Study
Brief Title: Cortisol Measurement During Intravenous Access With a Medical Clown
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0261-14-TLV
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2016-04

CONDITIONS: Stress, Physiological
Keywords: Medical clown; Pediatric emergency medicine
MeSH Terms: interventions — Laughter Therapy

ARMS (2):
- No clown (No Intervention): Routine venipuncture without distraction
- Clown (Active Comparator): A medical clown is present in the procedure room during venipuncture
  Interventions: Behavioral: Clown

INTERVENTIONS:
Behavioral: Clown — Comparison of routine venipuncture with a distraction technique by a medical clown
  Arms: Clown

SUMMARY:
The purpose of this study is to determine whether the presence of a medical clown in a pediatric emergency department procedure room would reduce children's anxiety. The investigators hypothesize that this positive influence will be expressed as lower levels of the stress hormone (Cortisol) in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing venous blood sampling or insertion of an intravenous canula
* Normal development according to parents

Exclusion Criteria:

* Critically ill children (e.g. shock, respiratory distress or failure)
* Children whose blood work or intravenous canula must be obtained rapidly for therapeutic reasons (e.g. antibiotic administration in a patient with severe bacterial infections)
* Known adrenal or pituitary disease
* Children who have received glucocorticoids during the preceeding six weeks

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Blood Cortisol level | During intravenous cannulation or blood sampling

SECONDARY OUTCOMES:
Vital signs (heart rate, respiratory rate, blood pressure) | During intravenous cannulation or blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Rimon, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Miguel Glatstein, MD, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel